CLINICAL TRIAL: NCT04481659
Title: Completely Abdominal Approach Laparoscopic Partial Intersphincteric Resection for Rectal Cancer: A Non-randomized, Prospective, Single-center Study
Brief Title: Completely Abdominal Approach Laparoscopic Partial Intersphincteric Resection for Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhongnanH1
Record Dates: First submitted 2020-07-19; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): Patients who are initially staged as T1-2, according to MRI and intraluminal ultrasound, are assigned to the direct surgery group (determined by the multidisciplnary team [MDT] group)
  Interventions: Procedure: Lap partial ISR
- B group (Experimental): Patients who are initially staged as T3M0, according to MRI and intraluminal ultrasound, should undertake preoperative chemoradiotherapy (determined by the MDT group). The operation was performed 8-12 weeks after the end of the chemoradiotherapy.
  Interventions: Combination Product: NCRT+Lap partial ISR

INTERVENTIONS:
Procedure: Lap partial ISR — A direct laparoscopic surgery with completely abdominal approach laparoscopic partial intersphincteric resection
  Arms: A group
Combination Product: NCRT+Lap partial ISR — Preoperative radiation and chemotherapy + laparoscopic completely abdominal approach laparoscopic partial intersphincteric resection
  Arms: B group

SUMMARY:
The conventional intersphincteric resection (ISR) for low rectal cancer requires a combined abdominal and perineal approach, and followed with a handsewn coloanal anastomosis, which is time consuming and difficult to accomplish. A complete laparoscopic abdominal approach partial intersphincteric resection has been proved to be a safe and feasible alternative for low rectal cancer treatment, with the advantages of technical convenience and avoiding a permanent ostomy. But there are few reports concerning differences in clinical outcomes between patients with or without neoadjuvant chemoradiotherapy undergoing partial ISR surgery. Therefore, it is necessary to compare the functional outcomes (including anal and sexual function, and postoperative quality of life [QOL]) and oncologic outcomes of patients who underwent completely abdominal approach laparoscopic partial ISR surgery after neoadjuvant chemoradiotherapy, with those who received ISR surgery directly. Furthermore, the operation difficulty between the above two groups is also worthy of intensive study.

DETAILED DESCRIPTION:
Patients with cT1 to cT2 low rectal cancer are directly operated through completely abdominal approach laparoscopic partial ISR surgery. Patients with cT3 low rectal cancer are firstly treated with standard neoadjuvant chemoradiotherapy until down staged to ycT1 to ycT2. The postoperatively functional outcomes and oncologic outcomes between the two groups are compared, including anal and sexual function, QOL and local recurrence rate. The operation difficulty between the above two groups is also investigated, including operation time, the intraoperative and postoperative complications, mesorectum integrity, time for mobilizing the intersphincteric plane, the intactness of the fascia of the levator ani muscle, pubis coccygeus, puborectalis, and external sphincter.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven moderate or well differentiated adenocarcinoma
* Rullier classification of low rectal cancer (types Ⅱ: juxta-anal tumor)
* Clinical staging: initially staged as T1 -2 or down staged to T1-2 after neoadjuvant chemoradiotherapy;

Exclusion Criteria:

* Without signing informed consent, poor compliance
* Unfit for laparoscopy
* Other serious diseases not suitable for participating in this clinical trial
* A degree of preoperative fecal incontinence
* After preoperative neoadjuvant chemoradiotherapy, the sphincter function, sexual function and others involved in this trail are seriously affected

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-19 (Estimated); Primary Completion 2025-07-19 (Estimated); Study Completion 2025-07-19 (Estimated)

PRIMARY OUTCOMES:
The damage degree of anal function | 5 years
  The value of this index in group A was defined as the preoperative anal function score minus the postoperative anal score. The value of this index in group B was defined as the anal function score which the patients have completed the standard neoadjuvant therapy minus the postoperative anal function score.

SECONDARY OUTCOMES:
Time for mobilizing the intersphincteric space | 5 years
  Time for mobilizing the intersphincteric space
The intactness of levator anus muscle fascia | 5 years
  The intactness of levator anus muscle fascia
he quality of specimen pathology: total mesorectal excision (TME) quality, the involvement of distal margin and circumferential margin | 5 years
  The quality of specimen pathology: total mesorectal excision (TME) quality, the involvement of distal margin and circumferential margin
Intraoperative and postoperative complications | 5 years
  Intraoperative and postoperative complications
Local recurrence | 5 years
  Local recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital, Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided